CLINICAL TRIAL: NCT01588457
Title: Sequential Multiple Assignment Randomized Treatment (SMART) for Bipolar Disorder
Brief Title: Sequential Multiple Assignment Treatment for Bipolar Disorder
Acronym: SMART
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC20110361H; 1P30MH086045-01A2 (NIH)
Record Dates: First submitted 2012-02-29; First posted 2012-05-01 (Estimated); Results first posted 2020-08-14 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Bipolar I Disorder; Bipolar II Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Lithium; Lithium Carbonate; Valproic Acid; Lamotrigine; Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Lithium (Active Comparator): This open methods advancement study will randomize BD patients with clinically significant symptoms to treatment with one of two mood stabilizers, lithium [Li] at baseline. Lithium is one of these two mood stabilizers. The person may or may not stay solely on lithium throughout the study.
  Interventions: Drug: Lithium
- Divalproex (Active Comparator): This open methods advancement study will randomize BD patients with clinically significant symptoms to treatment with one of two mood stabilizers, divalproex (DV)at baseline. Divalproex is one of these two mood stabilizers. The person may or may not stay solely on divalproex throughout the study.
  Interventions: Drug: Divalproex
- Lithium plus Quetiapine (Active Comparator): Those who develop protocol defined depression will then be randomized to a mood stabilizer (lithium) + quetiapine [QT].
  Interventions: Drug: Lithium; Drug: Quetiapine
- Lithium plus Lamotrigine (Active Comparator): Those who develop protocol defined depression will then be randomized to a mood stabilizer (lithium) + lamotrigine (LM).
  Interventions: Drug: Lithium; Drug: Lamotrigine
- Divalproex plus Quetiapine (Active Comparator): Those who develop protocol defined depression will then be randomized to a mood stabilizer (divalproex) + quetiapine [QT].
  Interventions: Drug: Divalproex; Drug: Quetiapine
- Divalproex plus Lamotrigine (Active Comparator): Those who develop protocol defined depression will then be randomized to a mood stabilizer (divalproex) + lamotrigine (LM).
  Interventions: Drug: Divalproex; Drug: Lamotrigine

INTERVENTIONS:
Drug: Lithium — Therapeutic dosage as indicated by participants condition with blood levels. LI will be dosed to attain Li of ≥0.5mEq/L (milliequivalents per liter).
  Other Names: Lithium Carbonate
  Arms: Lithium; Lithium plus Lamotrigine; Lithium plus Quetiapine
Drug: Divalproex — DV will be dosed to attain DV levels of ≥45mg/L.
  Other Names: Depakote; Depakote ER
  Arms: Divalproex; Divalproex plus Lamotrigine; Divalproex plus Quetiapine
Drug: Lamotrigine — LM will be incrementally dosed up to 400 mg/day, or, in combination with DV, 200 mg/day. Dosage may be reduced for adverse effects to one half of the target dose.
  Other Names: Lamictal
  Arms: Divalproex plus Lamotrigine; Lithium plus Lamotrigine
Drug: Quetiapine — QT will be started at 50 mg/day and titrated up to 300 mg as tolerated. QT will be discontinued if not tolerated at 100mg/day and the patient will be treated according to guidelines.
  Other Names: Seroquel
  Arms: Divalproex plus Quetiapine; Lithium plus Quetiapine

SUMMARY:
The purpose of this study is to compare which of the two mood stabilizers (drugs that help to steady/stabilize mood in patients with bipolar disorder (BD)), lithium and divalproex, is more effective in patients with bipolar disorder over 26 weeks. The study will also compare if lithium or divalproex used alone versus lithium or divalproex used with quetiapine versus lithium or divalproex used with lamotrigine is more effective when symptoms of depression develop.

DETAILED DESCRIPTION:
This open methods advancement study will randomize BD patients with clinically significant symptoms to treatment with one of two mood stabilizers (MS), lithium [Li] or divalproex [Div]. Those who develop protocol defined depression will then be randomized to a MS alone, MS + quetiapine [QTP] or MS + lamotrigine [LTG]. A SMART strategy employs a rule for adding new treatments based on each patient's current illness state and response during the trial, mimicking the adaptive nature of treatment selection which occurs in clinical settings, but in a controlled way which allows application of causal inference. By using early indices of response to dynamically alter treatment decisions to improve outcome, SMART eliminates unmeasured confounders associated with treatment decisions that are not randomized, as occurs in data mining exercises and in other non-randomized decisions in studies which randomize one variable at baseline. This sequential adaptive design represents a methodological innovation in bipolar trial history which will have particular implications for effectiveness studies.

Specific Aim A.1: Assess the feasibility of a SMART design in the conduct of an effectiveness study over 26 weeks in patients with BD (bipolar disorder).

Aim A.2 Compare the effectiveness of Li to Div as a primary component of treatment for BD over 26 weeks.

Aim A.3: Assess the effectiveness of MS + QTP and MS + LTG versus MS in subjects who develop depression.

A4. Exploratory Aims: 1.Determine the effects of ethnicity, language facility, education and stress as moderators of treatment outcomes; 2. Explore the use of novel statistical methodologies to more informatively characterize illness trajectories in response to the interventions. In the aggregate these aims also will clarify whether the SMART confirms results provided by traditional, single point randomized controlled trials (RCTs).

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV TR (Diagnostic and Statistical Manual Edition IV Text Revision) diagnosis BD I or II as assessed by MINI PLUS (Mini International Neuropsychiatric Interview PLUS)
* Male or female ≥ 18 years old
* Currently symptomatic with a CGI-BP-S ≥3 for mania/hypomania &/or depression for ≥ 2 weeks
* One of the following indicators of recent active illness: a depressive or manic or hypomanic or mixed episode in the past 12 months
* If female of child bearing age must use effective birth control.

Exclusion Criteria:

* Unwilling or unable to comply with study requirements
* Renal impairment (serum creatinine > 1.5 mg/dL)
* If maintained on thyroid medication must be euthyroid for at least 1 month before Visit 1
* Patients who have had intolerable side effects to QTP, Li, Div, or LTG
* Patients whose clinical status requires inpatient care
* Drug/alcohol dependence within the past 30 days
* Pregnancy as determined by serum pregnancy test or breastfeeding
* History of poor response to Li at a serum Li of ≥ 0.5 mEq/L (milliequivalents per Liter) or Div at a serum level of ≥ 45 mg/dL for at least 2 weeks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2011-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles L. Bowden, M.D., Principal Investigator — University of Texas; Joseph R Calabrese, M.D., Principal Investigator — Case Western Reserve University
Locations (2):
- United States (2):
  - Case Western Reserve University, Cleveland, Ohio
  - University of Texas Health Science Center, San Antonio, Texas

REFERENCES:
- [Derived] Hashimoto Y, Kotake K, Watanabe N, Fujiwara T, Sakamoto S. Lamotrigine in the maintenance treatment of bipolar disorder. Cochrane Database Syst Rev. 2021 Sep 15;9(9):CD013575. doi: 10.1002/14651858.CD013575.pub2. PMID 34523118

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After a washout period of up to 1 week, subjects will be openly randomized to treatment with Lithium (Li) or Divalproex (Div) for 2 weeks. Subjects who become intolerant to lithium or divalproex at any point will be crossed over to the other mood stabilizer and continued in the study, or terminate early.
Groups:
- Randomization to Lithium; Randomization to Divalproex: Subjects enrolled will be randomized to one of two mood stabilizers, Lithium (Li) or Divalproex (Div) in Randomization 1. If subjects show no symptoms, they will complete at the end of this phase of treatment.
- Monotherapy Li or Div Plus Quetiapine: Subjects who were on Li or Div and developed symptoms of depression had Quetiapine added to their treatment regimen
- Monotherapy Li or Div Plus Lamotrigine: Subjects who were on monotherapy Li or Div who developed symptoms of depression had Lamotrigine added to their regimen
Period: Randomization 1
Arm/Group | Randomization to Lithium | Randomization to Divalproex | Monotherapy Li or Div Plus Quetiapine | Monotherapy Li or Div Plus Lamotrigine
Started (Not all subjects were eligible to progress to from Randomization 1 to 2 based on depression symptoms) | 53 | 59 | 0 (No subject assigned during first randomization to monotherapy) | 0 (No subject assigned during first randomization to monotherapy)
Completed | 30 | 43 | 0 | 0
Not Completed | 23 | 16 | 0 | 0
Period: Randomization 2
Arm/Group | Randomization to Lithium | Randomization to Divalproex | Monotherapy Li or Div Plus Quetiapine | Monotherapy Li or Div Plus Lamotrigine
Started (Some subjects completed at the end of Randomization 1 and did not progress to randomization 2) | 21 (Some subjects who completed the first randomization had QTP or LTG added to regimen) | 31 (Some subjects who completed the first randomization had QTP or LTG added to regimen) | 17 (Assignment of Quetiapine plus monotherapy for symptoms of depression) | 18 (Assignment of Lamotrigine plus monotherapy for symptoms of depression)
Completed | 1 | 3 | 12 | 13
Not Completed | 20 | 28 | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Randomization to Divalproex: Subjects randomized to Divalproex at Randomization 1. Demographics were only tracked in the Randomization 1 phase.
- Randomization to Lithium: Subjects randomized to Lithium at Randomization 1. Demographics were only tracked in the Randomization 1 phase.
- Total: Total of all reporting groups
Arm/Group | Randomization to Divalproex | Randomization to Lithium | Total
Number analyzed (Participants) | 59 | 53 | 112
Age, Customized [Count of Participants; unit: Participants]
  Subjects over 18 years old | 59 | 53 | 112
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 32 | 69
  Male | 22 | 21 | 43
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Overall Total: African American | 8 | 7 | 15
  Overall Total: White (non Hispanic) | 33 | 26 | 59
  Overall Total: Hispanic | 15 | 19 | 34
  Overall Total: Asian/Asian American | 1 | 1 | 2
  Overall Total: Other | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 59 | 53 | 112

OUTCOME MEASURES:

1. Primary Outcome: Bipolar Inventory of Symptoms Scale (BISS)
Description: The BISS uses a structured interview to assess the full spectrum of symptoms associated with all primary clinical states in bipolar disorder, yielding a total severity, a depression, a mania, as well as dimensional scale scores. There are 42 items; each item is rated on a 0-4 scale. The BISS is a clinician-rated instrument. The Scale is rated as follows:
  0 Not at all
  1. Slight
  2. Mild
  3. Moderate
  4. Severe Each of the 42 items is rated separately, with a score, based on the most recent 7 day period. The mean score is calculated from the total score, giving an overall score out of 4, where 0 is slight and 4 is the most severe symptoms. A negative score indicated an improvement from baseline to 26 weeks.
Time Frame: Change from Baseline to 26 weeks
Measure: Mean (Standard Deviation); unit: calculated mean scale score
Groups:
- Divalproex After Randomization 1: After a washout period of up to 1 week, subjects will be openly randomized to treatment Divalproex for 2 weeks. Subjects who become intolerant to or divalproex at any point will be crossed over to the other mood stabilizer (Lithium) and continued in the study.
- Lithium After Randomization 1: After a washout period of up to 1 week, subjects will be openly randomized to treatment Lithium for 2 weeks. Subjects who become intolerant to or Lithium at any point will be crossed over to the other mood stabilizer (Divalproex) and continued in the study.
- Divalproex or Lithium Monotherapy: Group which continued monotherapy or divalproex after Randomization 2
- Lithium or Divalproex Plus Quetiapine: Group which had Quetiapine added to Lithium of Divalproex
- Lithium or Divalproex Plus Lamotrigine: Group which had Lamotrigine added to Lithium or Quetiapine
Arm/Group | Divalproex After Randomization 1 | Lithium After Randomization 1 | Divalproex or Lithium Monotherapy | Lithium or Divalproex Plus Quetiapine | Lithium or Divalproex Plus Lamotrigine
Number analyzed (Participants) | 59 | 53 | 17 | 17 | 18
calculated mean scale score
  Mania | -0.31 (NA) — Standard deviation is unavailable since the PI and statistician have retired and the information is unavailable. | -0.41 (NA) — Standard deviation is unavailable since the PI and statistician have retired and the information is unavailable. | 0.15 (NA) — Standard deviation is unavailable since the PI and statistician have retired and the information is unavailable. | -0.38 (NA) — Standard deviation is unavailable since the PI and statistician have retired and the information is unavailable. | -0.85 (NA) — Standard deviation is unavailable since the PI and statistician have retired and the information is unavailable.
  Depression | -0.71 (NA) — Standard deviation is unavailable since the PI and statistician have retired and the information is unavailable. | -0.20 (NA) — Standard deviation is unavailable since the PI and statistician have retired and the information is unavailable. | -0.18 (NA) — Standard deviation is unavailable since the PI and statistician have retired and the information is unavailable. | -0.61 (NA) — Standard deviation is unavailable since the PI and statistician have retired and the information is unavailable. | -0.95 (NA) — Standard deviation is unavailable since the PI and statistician have retired and the information is unavailable.
  Irritability | -0.50 (NA) — Standard deviation is unavailable since the PI and statistician have retired and the information is unavailable. | -0.39 (NA) — Standard deviation is unavailable since the PI and statistician have retired and the information is unavailable. | -0.27 (NA) — Standard deviation is unavailable since the PI and statistician have retired and the information is unavailable. | -0.66 (NA) — Standard deviation is unavailable since the PI and statistician have retired and the information is unavailable. | -0.96 (NA) — Standard deviation is unavailable since the PI and statistician have retired and the information is unavailable.
  Anxiety | -0.49 (NA) — Standard deviation is unavailable since the PI and statistician have retired and the information is unavailable. | -0.51 (NA) — Standard deviation is unavailable since the PI and statistician have retired and the information is unavailable. | 0.16 (NA) — Standard deviation is unavailable since the PI and statistician have retired and the information is unavailable. | -0.72 (NA) — Standard deviation is unavailable since the PI and statistician have retired and the information is unavailable. | -0.93 (NA) — Standard deviation is unavailable since the PI and statistician have retired and the information is unavailable.
  Psychosis | -0.14 (NA) — Standard deviation is unavailable since the PI and statistician have retired and the information is unavailable. | -0.25 (NA) — Standard deviation is unavailable since the PI and statistician have retired and the information is unavailable. | -0.27 (NA) — Standard deviation is unavailable since the PI and statistician have retired and the information is unavailable. | -0.14 (NA) — Standard deviation is unavailable since the PI and statistician have retired and the information is unavailable. | -0.16 (NA) — Standard deviation is unavailable since the PI and statistician have retired and the information is unavailable.

2. Secondary Outcome: Global Assessment of Functioning
Description: The Clinical Global Impression-Severity Scale (CGI-S) is used to assess global illness severity
  The CGI-S score change is measured from baseline to 26 weeks and is rated on a 7-point scale. The scale is read as follows:
  1. very much improved since the initiation of treatment
  2. much improved
  3. minimally improved
  4. no change from baseline (the initiation of treatment)
  5. minimally worse
  6. much worse
  7. very much worse since the initiation of treatment The score is calculated as a mean of all items, where 1 indicates improvement from inititation of visit, and 7 indicates the condition to be much worse since the inititation of treatment. A negative score indicates a change from worse to better.
Time Frame: Change from Baseline to 26 weeks
Measure: Mean (Standard Deviation); unit: calculated mean scale score
Groups:
- Divalproex After Randomization 1: After a washout period of up to 1 week, subjects will be openly randomized to Divalproex. Subjects who become intolerant to Divalproex at any point will be crossed over to the other mood stabilizer (Lithium) and continued in the study.
- Lithium After Randomization 1: After a washout period of up to 1 week, subjects will be openly randomized to Lithium. Subjects who become intolerant to or lithium at any point will be crossed over to the other mood stabilizer (divalproex) and continued in the study.
- Divalproex or Lithium Monotherapy: Group which continued monotherapy on Divalproex or Lithium
- Lithium or Divalproex Plus Quetiapine: Group which had Quetiapine added to Lithium or Divalproex
- Lithium or Divalproex Plus Lamotrigine: Group which had Lamotrigine added to Lithium or Divalproex
Arm/Group | Divalproex After Randomization 1 | Lithium After Randomization 1 | Divalproex or Lithium Monotherapy | Lithium or Divalproex Plus Quetiapine | Lithium or Divalproex Plus Lamotrigine
Number analyzed (Participants) | 59 | 53 | 17 | 17 | 18
calculated mean scale score
  CGI-Depression | -1.11 (NA) — PI and statistician have retired and do not have access to the data | -0.32 (NA) — PI and statistician have retired and do not have access to the data | -0.09 (NA) — PI and statistician have retired and do not have access to the data | -0.99 (NA) — PI and statistician have retired and do not have access to the data | -1.24 (NA) — PI and statistician have retired and do not have access to the data
  CGI-Mania | -0.69 (NA) — PI and statistician have retired and do not have access to the data | -1.12 (NA) — PI and statistician have retired and do not have access to the data | -0.19 (NA) — PI and statistician have retired and do not have access to the data | -0.71 (NA) — PI and statistician have retired and do not have access to the data | -1.81 (NA) — PI and statistician have retired and do not have access to the data
  CGI-Overall | -1.28 (NA) — PI and statistician have retired and do not have access to the data | -0.55 (NA) — PI and statistician have retired and do not have access to the data | -0.11 (NA) — PI and statistician have retired and do not have access to the data | -0.99 (NA) — PI and statistician have retired and do not have access to the data | -1.64 (NA) — PI and statistician have retired and do not have access to the data

3. Secondary Outcome: Baseline Randomization Percentage of Bipolar Types
Description: Percentages of Type I and Type II Bipolar Disorder included in Randomization groups
Time Frame: Baseline
Measure: Number; unit: percentage of participants
Groups:
- Bipolar Type 1 Divalproex Group; Bipolar Type 1 Lithium Group: Percentage of Bipolar Type 1 included in Randomization 1
- Bipolar Type II Divalproex Group; Bipolar Type II Lithium Group: Percentage of Bipolar Type II included in Randomization 1
Arm/Group | Bipolar Type 1 Divalproex Group | Bipolar Type II Divalproex Group | Bipolar Type 1 Lithium Group | Bipolar Type II Lithium Group
Number analyzed (Participants) | 59 | 53 | 59 | 53
percentage of participants | 70 | 74.1 | 30 | 25.9

4. Secondary Outcome: Demographic in Randomization 1 Group
Description: Baseline demographic percentages of subject randomized to either Divalproex or Lithium at the first randomization
Time Frame: Baseline
Measure: Number; unit: percentage of subjects
Groups:
- Divalproex: Subjects randomized to Divalproex at the first randomization
- Lithium: Subjects randomized to Lithium at the first randomization.
Arm/Group | Divalproex | Lithium
Number analyzed (Participants) | 59 | 53
percentage of subjects
  Single never married | 27.1 | 33.3
  Married | 55.9 | 37.0
  Disrupted Marriage | 17.0 | 29.6

ADVERSE EVENTS:
Description: Adverse events were only collected for Lithium and Divalproex interventions. Adverse events were not tracked for monotherapy plus QTP or LTG (in Randomization 2 of the study).
Groups:
- Divalproex: After a washout period of up to 1 week, subjects will be openly randomized to treatment Divalproex for 2 weeks. Subjects who become intolerant to or divalproex at any point will be crossed over to the other mood stabilizer (Lithium) and continued in the study. Adverse events were not collected for Randomization 2.
- Lithium: After a washout period of up to 1 week, subjects will be openly randomized to treatment Lithium for 2 weeks. Subjects who become intolerant to or Lithium at any point will be crossed over to the other mood stabilizer (Divalproex) and continued in the study. Adverse events were not collected for Randomization 2.
Arm/Group | Divalproex | Lithium
Serious Adverse Events (participants affected / at risk) | 1/59 | 1/53
Other Adverse Events (participants affected / at risk) | 19/59 | 15/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Divalproex (N=59) | Lithium (N=53)
Shortness of Breath (Cardiac disorders) | 1 (1) | 0 (0)
Neurological symptoms (Nervous system disorders) | 0 (0) | 1 (1) — Headache, drowsiness, thirst
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Divalproex (N=59) | Lithium (N=53)
Nausea and Vomiting (Gastrointestinal disorders) | 19 (19) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No